CLINICAL TRIAL: NCT02783014
Title: Case-control Study Investigating Central Mechanisms of Overactive Bladder in Adults With Parkinson's Disease and Overactive Bladder and Adults With Parkinson's Disease Only
Brief Title: Investigating Central Mechanisms of Overactive Bladder in Adults With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: EvergreenHealth (Other)
Responsible Party: Principal Investigator, Pinky Agarwal, MD, MD, FAAN, EvergreenHealth
Other Study IDs: PADB-2016-01
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Parkinson's Disease
Keywords: overactive bladder
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates the central mechanisms of Overactive Bladder (OAB) in Patients with Parkinson's Disease (PD).

The plan is to enroll 10 adults with Parkinson's disease and Overactive bladder (PD + OAB) and 10 adults with Parkinson's disease only (PD). Both groups will undergo fMRI (functional MRI).

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a physical problem that causes strong urges to urinate, frequent urination, and sometimes urinary incontinence (accidental loss of urine control) commonly in patients with Parkinson' disease (PD) severely impacting their quality of life.

Unfortunately OAB in adults with PD is difficult to treat. This is largely because the mechanisms underlying OAB in adults with PD are not known. Recent functional MRI (fMRI) studies suggest that certain areas of the brain have an important role in OAB. Blood oxygenation level dependent (BOLD) fMRI is an imaging technique in which neural activity of a region of the brain can be measured by fluctuation in the BOLD signal. It is hoped that the findings of this study will allow the development of new treatments for adults with Parkinson's disease and overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD by United Kingdom (UK) brain bank criteria.
* PD patients with and without OAB as per bladder questionnaire.
* No change in PD medications after screening, with no dose changes during the study, except that pro re nata (PRN) doses of carbidopa/levodopa will be allowed to address periodic worsening of parkinsonian symptoms.
* Patient willing and able to complete study questionnaires.
* Use of other medication that could influence bladder function, will be permitted as long as the dose is stable during the study.
* Patient expects to have valid health insurance for the duration of the study period.

Exclusion Criteria:

* Women who are breast-feeding, pregnant or have the potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures).
* Cognitive deficits that in the opinion of the investigator would interfere with the subject's ability to give informed consent or perform study testing.
* Evidence of Urinary Tract Infection (UTI) at screening.
* Bladder pain or history of chronic inflammation such as interstitial cystitis, recurrent UTIs, bladder stones, bladder obstruction, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs.
* Adults who have an interstim device in place.
* Claustrophobia, occupational risk for ferrous metal in the eye, or having an implantable medical device or foreign body precluding fMRI (e.g. cardiac pacemaker, metallic fragment, orthopedic hardware).
* Intravesical botulinum toxin treatment within the previous six months of screening.
* Use of indwelling catheter or self-catheterization.
* Any other serious and/or unstable medical condition

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 adults with Parkinson's disease (PD) and Overactive Bladder (OAB) and 10 adults with PD only.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Comparison of perfusion activity in the Limbic System | 1 hour functional Magnetic Resonance Imaging (fMRI)
  Comparison of the perfusion activity in the limbic system between subjects with Parkinson's Disease and Overactive Bladder and Parkinson's disease only using Blood Oxygenation Level Dependent (BOLD) functional Magnetic Resonance Imaging (fMRI) contrast maps. It will be performed at the second visit.

SECONDARY OUTCOMES:
Determination on the relationship of perfusion activity in the limbic system and anxiety. | 1 hour functional Magnetic Resonance Imaging (fMRI) - 10 Minutes questionnaire.
  Determination of the relationship of perfusion activity in the limbic system and anxiety scores (using Zung's Self-rating Anxiety Scale (SAS)) in subjects with Parkinson's Disease and Overactive Bladder.

CONTACTS AND LOCATIONS:
Overall Officials: Pinky Agarwal, MD, Principal Investigator — EvergreenHealth
Locations (1):
- EvergreenHealth, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley CS, Rovner ES, Morgan MA, Berlin M, Novi JM, Shea JA, Arya LA. A new questionnaire for urinary incontinence diagnosis in women: development and testing. Am J Obstet Gynecol. 2005 Jan;192(1):66-73. doi: 10.1016/j.ajog.2004.07.037. PMID 15672005
- [Background] Chao-Gan Y, Yu-Feng Z. DPARSF: A MATLAB Toolbox for "Pipeline" Data Analysis of Resting-State fMRI. Front Syst Neurosci. 2010 May 14;4:13. doi: 10.3389/fnsys.2010.00013. eCollection 2010. PMID 20577591
- [Background] Goetz CG, Poewe W, Rascol O, Sampaio C, Stebbins GT, Counsell C, Giladi N, Holloway RG, Moore CG, Wenning GK, Yahr MD, Seidl L; Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: status and recommendations. Mov Disord. 2004 Sep;19(9):1020-8. doi: 10.1002/mds.20213. PMID 15372591
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Jain S. Multi-organ autonomic dysfunction in Parkinson disease. Parkinsonism Relat Disord. 2011 Feb;17(2):77-83. doi: 10.1016/j.parkreldis.2010.08.022. Epub 2010 Sep 20. PMID 20851033
- [Background] Kilpatrick LA, Kutch JJ, Tillisch K, Naliboff BD, Labus JS, Jiang Z, Farmer MA, Apkarian AV, Mackey S, Martucci KT, Clauw DJ, Harris RE, Deutsch G, Ness TJ, Yang CC, Maravilla K, Mullins C, Mayer EA. Alterations in resting state oscillations and connectivity in sensory and motor networks in women with interstitial cystitis/painful bladder syndrome. J Urol. 2014 Sep;192(3):947-55. doi: 10.1016/j.juro.2014.03.093. Epub 2014 Mar 26. PMID 24681331
- [Background] McGrother CW, Jagger C, Clarke M, Castleden CM. Handicaps associated with incontinence: implications for management. J Epidemiol Community Health. 1990 Sep;44(3):246-8. doi: 10.1136/jech.44.3.246. PMID 2148771
- [Background] Nardos R, Gregory WT, Krisky C, Newell A, Nardos B, Schlaggar B, Fair DA. Examining mechanisms of brain control of bladder function with resting state functional connectivity MRI. Neurourol Urodyn. 2014 Jun;33(5):493-501. doi: 10.1002/nau.22458. Epub 2013 Jul 3. PMID 23908139
- [Background] Sakakibara R, Nakazawa K, Uchiyama T, Yoshiyama M, Yamanishi T, Hattori T. Micturition-related electrophysiological properties in the substantia nigra pars compacta and the ventral tegmental area in cats. Auton Neurosci. 2002 Nov 29;102(1-2):30-8. doi: 10.1016/s1566-0702(02)00180-7. PMID 12492133
- [Background] Sakakibara R, Panicker J, Finazzi-Agro E, Iacovelli V, Bruschini H; Parkinson's Disease Subcomittee, The Neurourology Promotion Committee in The International Continence Society. A guideline for the management of bladder dysfunction in Parkinson's disease and other gait disorders. Neurourol Urodyn. 2016 Jun;35(5):551-63. doi: 10.1002/nau.22764. Epub 2015 Mar 25. PMID 25810035
- [Background] Sakakibara R, Shinotoh H, Uchiyama T, Sakuma M, Kashiwado M, Yoshiyama M, Hattori T. Questionnaire-based assessment of pelvic organ dysfunction in Parkinson's disease. Auton Neurosci. 2001 Sep 17;92(1-2):76-85. doi: 10.1016/S1566-0702(01)00295-8. PMID 11570707
- [Background] Sakakibara R, Tateno F, Kishi M, Tsuyuzaki Y, Uchiyama T, Yamamoto T. Pathophysiology of bladder dysfunction in Parkinson's disease. Neurobiol Dis. 2012 Jun;46(3):565-71. doi: 10.1016/j.nbd.2011.10.002. Epub 2011 Oct 10. PMID 22015601
- [Background] Sakakibara R, Uchiyama T, Yamanishi T, Shirai K, Hattori T. Bladder and bowel dysfunction in Parkinson's disease. J Neural Transm (Vienna). 2008;115(3):443-60. doi: 10.1007/s00702-007-0855-9. Epub 2008 Mar 10. PMID 18327532
- [Background] Song XW, Dong ZY, Long XY, Li SF, Zuo XN, Zhu CZ, He Y, Yan CG, Zang YF. REST: a toolkit for resting-state functional magnetic resonance imaging data processing. PLoS One. 2011;6(9):e25031. doi: 10.1371/journal.pone.0025031. Epub 2011 Sep 20. PMID 21949842
- [Background] Uchiyama T, Sakakibara R, Hattori T, Yamanishi T. Short-term effect of a single levodopa dose on micturition disturbance in Parkinson's disease patients with the wearing-off phenomenon. Mov Disord. 2003 May;18(5):573-8. doi: 10.1002/mds.10403. PMID 12722172
- [Background] Valentino RJ, Wood SK, Wein AJ, Zderic SA. The bladder-brain connection: putative role of corticotropin-releasing factor. Nat Rev Urol. 2011 Jan;8(1):19-28. doi: 10.1038/nrurol.2010.203. Epub 2010 Dec 7. PMID 21135878
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928